CLINICAL TRIAL: NCT06998732
Title: Using Biased Coin Design (BCD) to Measure the ED95 of Remimazolam-Assisted Sedation in Arteriovenous Fistula Creation Surgery
Brief Title: BCD to Measure the ED95 of Remimazolam-Assisted Sedation in Arteriovenous Fistula Creation Surgery
Acronym: BCD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gang Chen (Other)
Responsible Party: Sponsor-Investigator, Gang Chen, chief physician, Sir Run Run Shaw Hospital
Organization: Sir Run Run Shaw Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: remimazolam; 13152 (Other Grant/Funding Number: Gang Chen)
Record Dates: First submitted 2025-05-14; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Uremia
Keywords: Biased Coin Design; uremia; remimazolam; ED95
MeSH Terms: conditions — Uremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- remimazolam group (Experimental): Measurement of ED95 in uremic patients sedated with remimazolam using the BCD method
  Interventions: Drug: remimazolam sedation

INTERVENTIONS:
Drug: remimazolam sedation — remimazolam sedation

SUMMARY:
This study intends to measure the ED95 of remimazolam-assisted sedation in arteriovenous fistula creation by BCD.

DETAILED DESCRIPTION:
Operative venous fistula (AVF) under local anaesthesia is a common surgical procedure for long-term haemodialysis patients. A common surgical procedure for patients with renal failure on dialysis. However, due to the long duration of the procedure, patients are prone to anxiety and nervousness that Especially if it is difficult to keep quiet during the operation, it may lead to blood pressure fluctuation and other complications, affecting the operation's smooth progress of the procedure. Moderate sedation is particularly important in this type of surgery, as it can effectively relieve the patient's tension and stabilise vital signs, It can effectively relieve the patient's tension, stabilise vital signs and reduce the patient's discomfort, thus contributing to the successful completion of the operation.This study intends to measure the ED95 of remazolam-assisted sedation in arteriovenous fistula creation by BCD. This will provide a scientific basis for anaesthetic drug selection in uremic patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old (including borderline values).
* Elective surgical patients under local anaesthesia for operation of AVF
* Voluntary participation in this study and signing of informed consent.
* American Society of Anesthesiologists (ASA) classification < Grade IV.
* BMI range: 18-28kg/m2 (including borderline values).

Exclusion Criteria:

* hypersensitivity to remimazolam or benzodiazepines.
* patients with severe cardiac, pulmonary, neurological diseases or liver failure. -- Preoperative use of sedative drugs, anticonvulsants, etc.
* patients who cannot cooperate with postoperative recovery or follow-up.
* vulnerable groups, including those with mental illness, cognitive impairment, critically ill patients, pregnant women, illiterates, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
ED95 | 1 day
  the dose of Remimazolam that provides satisfactory sedation in 95% of patients.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol